CLINICAL TRIAL: NCT01782365
Title: Impact of Transcranial Slow Oscillating Stimulation on Memory Consolidation During Slow Wave Sleep of a Daytime Nap in Patients With Mild Cognitive Impairment(MCI)
Brief Title: Effects of Brain Stimulation During a Daytime Nap on Memory Consolidation in Patients With Mild Cognitive Impairment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Agnes Flöel, Prof. Agnes Flöel, MD, Charite University, Berlin, Germany
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: Nap-tSOS-MCI
Record Dates: First submitted 2013-01-31; First posted 2013-02-01 (Estimated); Last update posted 2021-05-14 (Actual); Status verified 2021-05

CONDITIONS: Mild Cognitive Impairment, So Stated
Keywords: mild cognitive impairment; dementia; MCI; brain stimulation; tSOS; tDCS; sleep; nap; daytime sleep; memory; memory consolidation
MeSH Terms: conditions — Cognitive Dysfunction; Dementia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 0,75 Hz stimulation (Experimental): transcranial slow oscilliating stimulation (tSOS)during periods of SWS
  Interventions: Device: 0,75 Hz stimulation
- SHAM stimulation (Sham Comparator): SHAM stimulation during periods of SWS
  Interventions: Device: SHAM stimulation

INTERVENTIONS:
Device: SHAM stimulation — no stimulation
  Arms: SHAM stimulation
Device: 0,75 Hz stimulation
  Other Names: oscillating direct current brain stimulation
  Arms: 0,75 Hz stimulation

SUMMARY:
The beneficial effect of nocturnal as well as daytime sleep on memory consolidation is well-documented in young, healthy subjects. Slow wave sleep (SWS), in particular, with its slow oscillating activity have shown to enhance declarative, hippocampus-dependent memory representations. This impact of sleep on memory performance can be additionally enhanced by exogeneous induction of transcranial slow oscillating stimulation (tSOS) within the frequency range of SWS in humans (0,7- 0,8 Hz) during sleep, as has been demonstrated in young, healthy subjects. If patients with amnestic mild cognitive impairment (MCI)- usually characterized by initial difficulties in hippocampus dependent memory functions - benefit from transcranial slow oscillatory stimulation (tSOS) during sleep as well has not been studied so far. The primary goal of the study is therefore to investigate the impact of oscillating current stimulation (tSOS) during a daytime nap on declarative memory consolidation in MCI patients.

ELIGIBILITY:
Inclusion Criteria:

* amnestic and amnestic plus MCI-patients:

  1. Concern reflecting a change in cognition reported by patient or informant or clinician (i.e., historical or observed evidence of decline over time)
  2. Objective evidence of memory impairment; additional cognitive domains may be affected as well;
  3. Preservation of independence in functional abilities
  4. no dementia
* age: 50-90 years

Exclusion Criteria:

* untreated severe internal or psychiatric diseases
* epilepsy
* other severe neurological diseases eg., previous major stroke, brain tumour
* dementia
* contraindications to MRI

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2013-08-08 (Actual); Primary Completion 2016-04-26 (Actual); Study Completion 2016-08-30 (Actual)

PRIMARY OUTCOMES:
Retention of declarative memories after 0.75 Hz stimulation during SWS, vs after sham stimulation during SWS | 4 Weeks
  Retention between stimulation conditions (0.75 Hz during SWS, vs sham stimulation during SWS) in the declarative memory task.

SECONDARY OUTCOMES:
Amount of Slow wave Sleep, spindels, eeg-correlates, further memory systems | 4 Weeks
  1. Amount of slow wave sleep assessed by standard polysomnographic criteria in 0,75 Hz vs SHAM stimulation during SWS.
  2. Spindel activity during sleep indicated via several spindel parameters like number, duration, frequency of spindles; compared between 0,75 Hz and SHAM stimulation during SWS.
  3. Neuronal correlates (EEG-power in slow oscillation frequency bands induced by 0,75 Hz vs SHAM stimulation during SWS; EEG-correlates of encoding and retrieval of a declarative memory task).
  4. Performance in further memory systems (procedural), compared between 0,75 Hz and SHAM stimulation during SWS.

CONTACTS AND LOCATIONS:
Overall Officials: Agnes Flöel, Professor, Study Chair — Charite Universitätsmedizin Berlin - Neurologie
Locations (1):
- Charite CCM Neurologie Berlin, Berlin, Germany

REFERENCES:
- [Background] Marshall L, Helgadottir H, Molle M, Born J. Boosting slow oscillations during sleep potentiates memory. Nature. 2006 Nov 30;444(7119):610-3. doi: 10.1038/nature05278. Epub 2006 Nov 5. PMID 17086200
- [Background] Diekelmann S, Born J. The memory function of sleep. Nat Rev Neurosci. 2010 Feb;11(2):114-26. doi: 10.1038/nrn2762. Epub 2010 Jan 4. PMID 20046194
- [Background] Ferrucci R, Mameli F, Guidi I, Mrakic-Sposta S, Vergari M, Marceglia S, Cogiamanian F, Barbieri S, Scarpini E, Priori A. Transcranial direct current stimulation improves recognition memory in Alzheimer disease. Neurology. 2008 Aug 12;71(7):493-8. doi: 10.1212/01.wnl.0000317060.43722.a3. Epub 2008 Jun 4. PMID 18525028
- [Background] Naismith SL, Lewis SJ, Rogers NL. Sleep-wake changes and cognition in neurodegenerative disease. Prog Brain Res. 2011;190:21-52. doi: 10.1016/B978-0-444-53817-8.00002-5. PMID 21531243
- [Background] Mednick SC, Cai DJ, Kanady J, Drummond SP. Comparing the benefits of caffeine, naps and placebo on verbal, motor and perceptual memory. Behav Brain Res. 2008 Nov 3;193(1):79-86. doi: 10.1016/j.bbr.2008.04.028. Epub 2008 May 8. PMID 18554731
- [Background] Mander BA, Santhanam S, Saletin JM, Walker MP. Wake deterioration and sleep restoration of human learning. Curr Biol. 2011 Mar 8;21(5):R183-4. doi: 10.1016/j.cub.2011.01.019. No abstract available. PMID 21377092
- [Background] Mednick S, Nakayama K, Stickgold R. Sleep-dependent learning: a nap is as good as a night. Nat Neurosci. 2003 Jul;6(7):697-8. doi: 10.1038/nn1078. PMID 12819785
- [Result] Ladenbauer J, Ladenbauer J, Kulzow N, de Boor R, Avramova E, Grittner U, Floel A. Promoting Sleep Oscillations and Their Functional Coupling by Transcranial Stimulation Enhances Memory Consolidation in Mild Cognitive Impairment. J Neurosci. 2017 Jul 26;37(30):7111-7124. doi: 10.1523/JNEUROSCI.0260-17.2017. Epub 2017 Jun 21. PMID 28637840
- [Derived] Rackoll T, Neumann K, Passmann S, Grittner U, Kulzow N, Ladenbauer J, Floel A. Applying time series analyses on continuous accelerometry data-A clinical example in older adults with and without cognitive impairment. PLoS One. 2021 May 13;16(5):e0251544. doi: 10.1371/journal.pone.0251544. eCollection 2021. PMID 33984029
- [Derived] Ladenbauer J, Ladenbauer J, Kulzow N, Floel A. Memory-relevant nap sleep physiology in healthy and pathological aging. Sleep. 2021 Jul 9;44(7):zsab002. doi: 10.1093/sleep/zsab002. PMID 33406266